CLINICAL TRIAL: NCT06913478
Title: Evaluation Of Effect of Axial Length on Cup-To-Disc Ratio Among Non- Glaucomatous Hypertensive Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/802
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Hypertensive Complication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational cross-sectional study aims to compare the effect of axial length on the cup-to-disc ratio in non-glaucomatous hypertensive patients. Data will be collected from Khursheed Begum Eye Hospital and LRBT Hospital, with a sample size of 104 participants. A purposive sampling technique will be used.

DETAILED DESCRIPTION:
Patients aged 18-70 years with systemic hypertension for at least one year and normal intraocular pressure will be included. Exclusion criteria include glaucoma, high myopia, hyperopia, ocular surgery, trauma, and optic nerve diseases. Axial length will be measured using optical biometry or A-scan ultrasonography, while the cup-to-disc ratio will be assessed through fundus examination using a slit lamp biomicroscope with a +90D lens or optical coherence tomography (OCT). Data will be meticulously documented, including patient demographics and medical history. The study will be completed within six months after approval, ensuring accurate and standardized measurements for reliable results.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with systemic hypertension for at least 1 year.
* Age between 18-70 years.
* Normal intraocular pressure (IOP<-21mmhg)
* Axial length between 21mm and 26mm (to exclude extreme refractive errors)

Exclusion Criteria:

* History of glaucoma or ocular hypertension.
* High myopia (<-6.00 D) or hyperopia (>+6.00D).
* History of ocular surgery, trauma, or retinal diseases.
* Any optic nerve diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: his observational cross-sectional study aims to compare the effect of axial length on the cup-to-disc ratio in non-glaucomatous hypertensive patients. Data will be collected from Khursheed Begum Eye Hospital and LRBT Hospital
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Axial length measured by biometry and CD ratio by slitlamp | 12 Months
  The axial length, measured in millimeters, is defined as the distance from the anterior surface of the cornea to the retinal pigment epithelium. The axial length can be measured using either ultrasound biometry (accomplished via direct contact or immersion) or optical biometry

CONTACTS AND LOCATIONS:
Locations (1):
- Alshifa eye clinic Ali Pur chattha, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No